CLINICAL TRIAL: NCT05753293
Title: Effect of Selected Types of Breathing Exercises on Different Outcome Measures in Covid-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basma Mosaad Abd-elrahman Abushady (Other)
Responsible Party: Sponsor-Investigator, Basma Mosaad Abd-elrahman Abushady, Master student at Department of Physical Therapy for Cardiovascular, Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P.T.REC/012/004298
Record Dates: First submitted 2023-02-24; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Sixty patients of both genders with age range from 40-50 years old will be recruited from El Khankah Centeral Hospital with positive nasopharyngeal swab samples and presence of ground-glass opacification in their chest computed tomography scan (CT-scan) will be assigned randomly into two groups A & B and take their medications.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bhastrika pranayama (Experimental): done in sitting posture and the following instructions: The back must be kept straight and shoulder muscles should be kept relaxed, patient was asked to close the right nostril with right thumb and to bring right elbow to the level of right shoulder.
  To close the eyes, inhale and exhale through left nostril-first slowly, then a little faster, The subject was asked to do the above steps about 20-25 times, (Then the subject was asked to take a long breath in and retain it for as long as possible, This is one cycle of Bhastrika pranayama. The subject has to repeat this cycle by closing left nostril and breathing through right nostril.
  Interventions: Other: breathing exercise
- Buteyko breathing exercise (Experimental): Step 1 beginning control pause (CP) the patient inhales and then exhales through the nose and then holds their breath until the point they feel either the first clear and distinct desire to breath or involuntary movement or jerk coming from diaphragm.Step 2 three to five minutes of relaxed reduced-volume breathing or slow breathing the patient gradually reduced their breathing until they feel a light lack of air. they sustain these while staying relaxed.
  Step 3 maximum pause (MP) the maximum pause begins with gentel inhalation and exhalation. Then the breath is held as long as possible but not to the point of severe discomfort.
  Step 2 and step 3 are then repeated up to 5 times. Final control pause: same as step 1.
  Interventions: Other: breathing exercise

INTERVENTIONS:
Other: breathing exercise — Buteyko breathing technique developed to control hyperventilation and anxiety which leads to shortness of breath. It uses series of exercises to teach patients to breathe less deeply and less rapidly /Bhastrika "Bellow Breathing" is diaphragmatic breathing - deep breathing involving the diaphragm rather than the accessory muscles. Regulated pranayama exercises require inhalation, maintaining isometric contraction of respiratory muscles and forceful expiration. These techniques will strengthen respiratory muscles
  Other Names: Bhastrika pranayama . Buteyko breathing exercise

SUMMARY:
Coronavirus disease 2019 (COVID-19) infection leads to significant respiratory that have negative impact on function and quality of life (QoL). Breathing exercises are effective and important in patients with COVID-19.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) infection leads to significant respiratory symptoms that have negative impact on function and quality of life (QoL). Breathing exercises are effective and important in patients with COVID-19.

This study aimed to evaluate the effect of Buteyko breathing versus Bhastrika Pranayama on different outcome measures in COVID-19 Patients.

Sixty patients of both genders with age range from 40-50 years old were recruited from El Khankah Centeral Hospital with positive nasopharyngeal swab samples and presence of ground-glass opacification in their chest computed tomography scan (CT-scan). Patients were assigned randomly into two groups A & B and took their medications. Group A received traditional physical therapy program (mobility exercises and Postural drainage) with Bhastrika Pranayama breathing exercise. Group B received traditional physical therapy program with Buteyko breathing exercise. Patients were assessed by Modified Borg Dyspnea Scale (MBS), blood samples (levels of CRP and d-dimer), six-minute walk test (6MWT), Pittsburgh Sleep Quality Index (PSQI), 36-Item Short-Form Health Survey (SF-36) Questionnaire.

ELIGIBILITY:
Inclusion criteria:

* Their age ranged from 40 to 50years old.
* with confirmed COVID-19 by positive nasopharyngeal swab samples and presence of ground-glass opacification in their chest computed tomography scan (CT-scan).
* Moderate hospitalized covid-19 patient.
* full consciousness and oriented.
* BMI 20-25 kg/m2.

Exclusion criteria:

* presence of any type of musculoskeletal disorder prohibits the patient from participating in the study
* history of chronic diseases as (diabetes, hypertension and heart diseases)
* Any type of obvious clinically mental or cognitive impairment.
* History of previous other respiratory disease.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Modified Borg Scale to Measure dyspnea: | week
  is a 0 to 10 rated numerical score used to measure dyspnea as reported by the patient with higher score indicates breathing problem.
Blood Samples: | week
  The blood samples will be collected before starting and at the end of the study to measure levels of CRP, d-dimer and CBC to test.
The Six-minute walk test: | week
  The six-minute walk test (6MWT) will be done pre & post exercise program.
Pittsburgh Sleep Quality Index (PSQI) | week
  The PSQI questionnaire was used to measure sleep quality using an 18-item scale containing seven items that included sleep quality, sleep duration, sleep latency, habitual sleep efficiency, sleep disturbance, use of sleeping medications, and daytime dysfunction. Each dimension scored between 0-3, with a total score ranging from 0-21, and a higher score indicating lower sleep quality
The 36-Item Short-Form Health Survey (SF-36) Questionnaire | week
  The SF-36 is a 36-item scale, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items) the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No